CLINICAL TRIAL: NCT01078025
Title: Evaluation of Microbial Colonisation and Contamination Caused by the Transvaginal and Transabdominal Access for Cholecystectomy
Acronym: NOBACT
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Andreas Zerz, MD, Cantonal Hospital St.Gallen, Departement of Surgery
Other Study IDs: EKSG09/150/1B
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-07

CONDITIONS: Cholecystectomy
Keywords: transvaginal access for cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- transvaginal hybrid cholecystectomy
  Interventions: Procedure: Smear test vaginally, intraabdominally
- laparoscopic cholecystectomy
  Interventions: Procedure: Smear test vaginally, intraabdominally

INTERVENTIONS:
Procedure: Smear test vaginally, intraabdominally — Pre- and intraoperative smear tests of the vagina and douglas are performed.
  Groups: transvaginal hybrid cholecystectomy
Procedure: Smear test vaginally, intraabdominally — Pre- and intraoperative smear tests of the vagina and douglas are performed.
  Groups: laparoscopic cholecystectomy

SUMMARY:
Transvaginal hybrid procedures are of interest as an available NOTES procedure for the clinical routine. The gynaecologists' experiences and the available studies report on low morbidity related to the transvaginal access. However, little is known about the vaginal and intraabdominal microbial contamination due to the transvaginal approach.

The aim of this cohort study is to evaluate the microbial colonisation and contamination in patients with transvaginal hybrid and conventional laparoscopic cholecystectomy.

Therefore, pre- and intraoperative microbiological evaluations will be performed in patients with transvaginal hybrid cholecystectomy and laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* indication for elective cholecystectomy
* informed consent for laparoscopic cholecystectomy or transvaginal hybrid cholecystectomy

Exclusion Criteria:

* cholecystitis
* intraabdominal infection
* existing antibiotic therapy
* adnexitis
* pelvic inflammatory disease
* infection (CRP > 10 mg /l; Lc > 11 G/l)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with symptomatic cholecystolithiasis and given informed consent for laparoscopic cholecystectomy or transvaginal hybrid cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Microbial colonisation and contamination vaginally and intraabdominally | 1 day

SECONDARY OUTCOMES:
Morbidity (wound, vaginal and intraabdominal infection) two weeks and six weeks postoperatively | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Zerz, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Department of Surgery, Sankt Gallen, St.Gallen, Switzerland